CLINICAL TRIAL: NCT00991354
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of PENNVAX™-B (Gag, Pol, Env) Vaccine, With or Without IL-12 DNA Plasmid, Delivered Via Electroporation in Healthy, HIV-1-Uninfected Adult Participants
Brief Title: Safety of and Immune Response to the PENNVAX-B DNA Vaccine With and Without IL-12 in HIV-uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 080; 10741 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Participants will receive 3 mg of PENNVAX-B vaccine or placebo at Months 0, 1, and 3.
  Interventions: Biological: PENNVAX-B
- Group 2 (Experimental): Participants will receive 3 mg of PENNVAX-B vaccine and 1 mg of IL-12 vaccine or placebo at Months 0, 1, and 3.
  Interventions: Biological: PENNVAX-B; Biological: IL-12 DNA plasmids
- Group 3 (Experimental): Participants will receive 3 mg of PENNVAX-B vaccine and 1 mg of IL-12 vaccine or placebo at Months 0, 1, and 3.
  Interventions: Biological: PENNVAX-B; Biological: IL-12 DNA plasmids

INTERVENTIONS:
Biological: PENNVAX-B — DNA vaccine encoding the Gag, Pol, and Env proteins of HIV
Biological: IL-12 DNA plasmids — Adjuvant for HIV vaccines
  Arms: Group 2; Group 3

SUMMARY:
An effective vaccine may be the only way to stop the HIV pandemic. The purpose of this study is to determine the safety of and immune response to the DNA vaccine, PENNVAX-B with or without an IL-12 adjuvant when given using electroporation.

DETAILED DESCRIPTION:
An effective and safe vaccine must be developed in order to halt the HIV pandemic. The purpose of this study is to assess the safety and immune response to the HIV DNA vaccine, PENNVAX-B when given with and without an IL-12 adjuvant and delivered via electroporation.

Participants in this study will be randomly assigned to one of three groups and will visit the study clinic 9 times over 9 months. Group 1 will enroll first. Participants in this group will receive 3 mg of the PENNVAX-B or placebo vaccine at Months 0, 1, and 3. Once safety data has been examined for Group 1, Group 2 will begin enrollment. Group 2 participants will receive 3 mg of PENNVAX-B vaccine plus 1 mg of IL-12 adjuvant or placebo at Months 0, 1, and 3. Once Group 1 and Group 2 safety data have been collected Group 3 will begin enrollment. These participants will also receive 3 mg of PENNVAX-B vaccine plus 1 mg of IL-12 adjuvant or placebo at Months 0, 1, and 3.

At clinic visits participants will have physical exams and blood and urine collected. After receiving study injections, participants will be observed in the clinic for at least 30 minutes. In addition, participants will be asked to monitor symptoms for 3 days after each injection.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study and the Step Study results; completes a questionnaire prior to first vaccination, with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Assessed by the clinic staff as being at "low risk" for HIV infection on the basis of behaviors within the 12 months prior to enrollment
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Certain laboratory values. Details on this criterion can be found in the protocol.
* Negative HIV-1 and -2 blood test: US participants must have a negative FDA-approved enzyme immunoassay (EIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Reproductive status: A volunteer who was born female must agree to consistently use effective contraception from at least 21 days prior to enrollment through the last required protocol clinic visit for sexual activity that could lead to pregnancy, or not be of reproductive potential, or be sexually abstinent
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion criteria:

* Within the 12 months prior to enrollment: excessive daily alcohol use or frequent binge drinking or chronic marijuana abuse or any other illicit drug use
* Within the 12 months prior to enrollment: a history of newly acquired or diagnosed syphilis; newly acquired gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, or chancroid
* Untreated or incompletely treated syphilis infection
* HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, documentation of the identity of the study control/placebo must be provided to the HVTN 080 PSRT, who will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA or for those who have received control/placebo in an experimental vaccine trial.
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray for allergic rhinitis; [2] topical corticosteroids for mild, uncomplicated dermatitis or [3] oral/parenteral corticosteroids given for non-chronic conditions not expected to recur [length of therapy 10 days or less with completion at least 30 days prior to enrollment])
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 60 days before first vaccination
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 080 study
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, Hepatitis A or B, HPV)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Allergy to amide-type local anesthetics
* Presence of implanted electronic medical device (e.g., pacemaker, implantable cardioverter defibrillator)
* A history of cardiac arrhythmia, e.g., supraventricular tachycardia, atrial fibrillation, or frequent ectopy on exam. (Not excluded: sinus arrhythmia)
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
* Autoimmune disease
* Immunodeficiency
* Asthma other than mild, well-controlled asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Angioedema within the last 3 years if episodes are considered serious or have required medication within the last 2 years
* Hypertension
* BMI > 30 kg/m2
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: a participant with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study.)
* Seizure disorder
* Asplenia: any condition resulting in the absence of a functional spleen
* Psychiatric condition that precludes compliance with the protocol
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of local injection/EP site reactogenicity signs and symptoms | Throughout study
Magnitude of local injection/EP site pain as measured by a VAS | Throughout study
Frequency of AEs categorized by MedDRA body system, MedDRA preferred term, severity and assessed relationship to study products; detailed description of all AEs meeting DAIDS criteria for expedited reporting | Throughout study
WBC, neutrophils, lymphocytes, hemoglobin, alkaline phosphatase, platelets, ALT, AST, creatinine, and creatine phosphokinase (CPK) | At baseline and post-vaccinations
Number of participants with early discontinuation of vaccinations and reason for discontinuation | Throughout study
Distribution of responses to questions regarding acceptability of study injections via EP | Throughout study

SECONDARY OUTCOMES:
Frequency of T-cell responses as measured by IFN-γ ELISpot | Two Weeks after the second and third vaccinations
Frequency of CD4+ T cell responses measured by intracellular cytokine staining (ICS) for IFN-γ and/or IL-2 to HIV potential T-cell epitope (PTE) peptide pools representing Gag, Pol, and Env | After the second and third vaccinations
Frequency of CD8+ T cell responses measured by ICS for IFN-γ and/or IL-2 to HIV PTE peptide pools representing Gag, Pol, and Env | After the second and third vaccinations
Frequency of humoral responses detected by HIV-1-specific neutralizing and binding antibody assays from serum samples | Two weeks after last vaccination
Frequency of vaccine-induced positive results with end-of-study HIV serological testing by commercial assays | Throughout study

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - 3535 Market Street CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine CRS, Nashville, Tennessee

REFERENCES:
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067